CLINICAL TRIAL: NCT03808402
Title: The Effect of Surfactant Dose on Outcomes in Preterm Infants With Respiratory Distress Syndrome
Brief Title: The Effect of Surfactant Dose on Outcomes in Preterm Infants With RDS
Acronym: OPTI-SURF
Status: Completed | Type: Observational
Sponsor: Chiesi UK (Industry)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 237111; 36652 (Other: CPMS)
Record Dates: First submitted 2019-01-14; First posted 2019-01-17 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Distress Syndrome; Bronchopulmonary Dysplasia
Keywords: Surfactant; Less Invasive Surfactant Administration; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High dose surfactant: Infants who receive a first dose of surfactant between 170 and 200 mg/kg
- Low dose surfactant: Infants who receive a first dose of surfactant between 100 and 130 mg/kg

SUMMARY:
A prospective observational study using de-identified data from the Neonatal Network Research Database (NNRD) supplemented by additional information on dose, method of surfactant administration and dosing frequency to assess whether the dose and method of administration of surfactant given to preterm infants with respiratory distress syndrome (RDS) affects neonatal outcomes.

DETAILED DESCRIPTION:
The rationale for this study is the clinical relevance of understanding whether surfactant dose affects neonatal outcomes in infants with RDS who are treated in the immediate postnatal period.

In a research environment, the dose of surfactant is rigorously controlled, usually administered at a dose of 100mg/kg or 200mg/kg. In clinical practice, clinicians more frequently follow the 'whole vial dosing' approach, where a full vial is given aiming to get as close as possible to the desired dose. Reasons for whole vial use include reduction of waste and administration of surfactant shortly after birth where an infant's weight is unknown. It is unclear whether whole vial dosing leads to under-dosing or over-dosing and whether either situation affects outcomes.

Information regarding the dose of surfactant delivered, and the method of administration, are not currently routinely recorded in the UK.

The primary objective of the study is to compare two dosing groups (100-130 mg/kg and 170-200 mg/kg) in terms of the proportions of infants who require mechanical ventilation within four days of birth.

ELIGIBILITY:
Inclusion Criteria:

* <37 weeks gestational age Requiring surfactant for Respiratory Distress Syndrome Record of birth weight available Born after study initiation

Exclusion Criteria:

* 37 weeks gestation age or above Parental opt-out

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborn infants born in neonatal units in the UK
Sampling Method: Non-Probability Sample
Enrollment: 2973 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Need for mechanical ventilation | Day 3 to 4 of life
  Survival without mechanical ventilation (excluding days 1 and 2 of life)

SECONDARY OUTCOMES:
Survival | To study completion, an average of 2 years
Number of doses of surfactant | To study completion, an average of 2 years
Total cumulative dose of surfactant (excluding the first dose) | To study completion, an average of 2 years
Survival with no respiratory support | On postnatal day 28
Survival with no respiratory support | 36 weeks gestation
Survival with no oxygen requirement | To study completion, an average of 2 years
Duration of mechanical ventilation (days) | To study completion, an average of 2 years
Duration of respiratory support (days) | To study completion, an average of 2 years
Two-year developmental outcomes | Two years
  As measured by Bailey's Score
Two-year developmental outcomes | Two years
  As measured by Composite Developmental Assessment

OTHER OUTCOMES:
Effect of dose on need for mechanical ventilation on days 3 and 4 (excluding days 1 and 2) | Day 3 to 4 of life
Effect of method of administration on need for mechanical ventilation on days 3 and 4 (excluding days 1 and 2) | Day 3 to 4 of life

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Goss, MBBS, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (29):
- United Kingdom (29):
  - William Harvey Hospital, Ashford, Kent
  - Birmingham Women's Hospital, Birmingham
  - Birmigham Heartlands Hospital, Birmingham
  - Royal Bolton Hospital, Bolton
  - Bradford Royal Infirmary, Bradford
  - Burnley General Hospital, Burnley
  - The Rosie Hospital, Cambridge
  - St Peter's Hospital, Chertsey
  - University Hospital Coventry, Coventry
  - Hull Royal Infirmary, Hull
  - Leeds General Infirmary, Leeds
  - Leicester Royal Infirmary, Leicester
  - Liverpool Women's Hospital, Liverpool
  - Homerton Hospital, London
  - University College Hospital, London
  - Guy's and St Thomas' Hospital, London
  - Chelsea and Westminster Hospital, London
  - St Mary's Hospital, Manchester
  - Wythenshawe Hospital, Manchester
  - The James Cook Hospital, Middlesbrough
  - University Hospital of North Tees, Middlesbrough
  - Royal Victoria Infirmary, Newcastle
  - Norfolk and Norwich University Hospital, Norwich
  - Queens Medical Centre, Nottingham
  - Royal Oldham Hospital, Oldham
  - John Radcliffe Hospital, Oxford
  - Queen Alexandra Hospital, Portsmouth
  - Jessop Wing, Sheffield
  - Princess Anne Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Goss KCW, Gale C, Malone R, Longford N, Ratcliffe K, Modi N. Effect of surfactant dose on outcomes in preterm infants with respiratory distress syndrome: the OPTI-SURF study protocol. BMJ Open. 2020 Dec 12;10(12):e038959. doi: 10.1136/bmjopen-2020-038959. PMID 33310795
- See also: Study website — https://www.leedsth.nhs.uk/research/clinical-trials/optisurf/